CLINICAL TRIAL: NCT05829330
Title: Ambulatory Versus Inpatient Initiation of Home Non-invasive Mechanical Ventilation in Patient With Amyotrophic Lateral Sclerosis: a Prospective, Noninferiority Randomized Controlled Trial (The NIB-study)
Brief Title: Ambulatory Versus Inpatient Initiation of Home Mechanical Ventilation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anne Kathrine Staehr-Rye (Other)
Responsible Party: Sponsor-Investigator, Anne Kathrine Staehr-Rye, M.D., Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-23005093
Record Dates: First submitted 2023-03-15; First posted 2023-04-25 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Hospitalization

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Outpatient (Active Comparator): Outpatient initiation of non-invasive mechanical ventilation
  Interventions: Other: Outpatient
- Hospitalization (Placebo Comparator): Initiation of non-invasive mechanical ventilation during hospitalization
  Interventions: Other: Hospitalization

INTERVENTIONS:
Other: Outpatient — Outpatient Initiation of noninvasive mechanical ventilation
  Arms: Outpatient
Other: Hospitalization — Initiation of non-invasive mechanical ventilation during hospitalization
  Arms: Hospitalization

SUMMARY:
The purpose of this investigation is to see if outpatient initiation of noninvasive home mechanical ventilation combined with closed telemonitoring and follow-up in patients with amyotrophic lateral sclerosis is non-inferior to initiation during admission to the hospital

The primary hypothesis is that outpatient intiation of noninvasive home mechanical ventilation combined with closed telemonitoring and follow-up is non-inferior to initiation during hospitalization in patients with amyotrophic lateral sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Diagnosed with amyotrophic lateral sclerosis
* Indication for start of non-invasive mechanical ventilation

Exclusion Criteria:

* No informed consent
* Does not understand Danish or English
* Indication for invasive mechanical ventilation
* No morning baseline PCO2
* Hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Use of non-invasive mechanical ventilation | The 83th to the 90th day after initiation of non-invasive mechanical ventilation
  Use of non-invasive mechanical ventilation in minutes per day

SECONDARY OUTCOMES:
Patient satisfaction with the treatment | Measured at the 3 months follow-up visit
  Patient satisfaction with the non-invasive mechanical ventilation (verbal-rating-score 1-5)
Patient satisfaction with the proces in relation to the start of the treatment | Measured at the 3 months follow-up visit
  Patient satisfaction with the proces in relation to the start of non-invasive mechanical ventilation (verbal-rating-score 1-5)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesia, Pain and REspiratory Support, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No